CLINICAL TRIAL: NCT01187914
Title: RADAR: Effect of Structural Remodeling on Scar Formation as Assessed by DE-MRI of the Left Atrium Following Open-Irrigation Cooled-Tip Radiofrequency Catheter Ablation of Paroxysmal Atrial Fibrillation
Brief Title: Effect of Structural Remodeling on Scar Formation as Assessed by DE-MRI of the Left Atrium
Acronym: RADAR
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Nassir F. Marrouche, MD, Associate Professor of cardiology, University of Utah
Other Study IDs: IRB_00042859
Record Dates: First submitted 2010-08-03; First posted 2010-08-24 (Estimated); Results first posted 2012-01-10 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Atrial Fibrillation
Keywords: Paroxysmal Atrial Fibrillation; Radio-frequency Ablation; Ablation; Open irrigation cooled-tip
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Open Irrigation: Those individuals who had an ablation using open irrigation cooled-tip RF ablation.

SUMMARY:
The purpose of this study is to evaluate the impact of pre-ablation fibrosis on scar formation in the left atrium of the heart. This will be assessed by delayed enhancement magnetic resonance imaging and will be looked at in patients who have undergone successful open irrigated cooled-tipped radio-frequency ablation of paroxysmal atrial fibrillation. Follow-up after ablation will be for 12 months.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is an electrophysiological condition characterized by disorganized electrical activity that involves the entire atria. AF manifests initially as paroxysms of arrhythmia that later progress into persistent and permanent forms. It is a progressive disease associated with structural, electrical and contractile changes in the left atrium (LA). A major determinant of the progression of AF is structural remodeling or fibrosis that occurs in the left atrium. A more extensively remodeled atrium presents the substrate needed for the arrhythmia to persist. Structural remodeling is also a major determinant for success of rhythm control strategies in AF. While catheter ablation has reproducibly been shown to be superior to anti-arrhythmic drug (AAD) therapy for rhythm control in AF, the success of this procedure is significantly affected by the extent of structural remodeling present at the time of catheter ablation.

Delayed-Enhancement Magnetic Resonance Imaging (DE-MRI) has been demonstrated to be a very effective modality in identifying fibrotic and scarred cardiac tissue with excellent correlation to electro-anatomical mapping. This is related to the characteristics of Gadolinium, an extracellular contrast agent that is very effective in identifying regions of fibrotic non-viable myocardium. DE-MRI technology can be a very powerful, non-invasive method, of identifying the extent and the distribution of structural remodeling or fibrosis associated with AF. Specific image acquisition sequences have allowed for reproducible identification of high pixel intensity regions within the 2-dimensional images of the atrial wall. 3-Dimensional reconstruction of the entire left atrium then provides a quantification of the overall volume occupied by these hyper-enhanced regions relative to the entire left atrial wall volume. Used prior to catheter ablation, DE-MRI can therefore identify regions of significant structural remodeling or fibrosis. The same technology has also been shown to be very useful in examining the amount and distribution of ablation-induced scarring.

Catheter ablation has emerged as an effective interventional therapeutic modality for AF patients. Current ablation techniques, including pulmonary vein antrum isolation (PVAI), use radiofrequency (RF) energy to induce thermal damage to the LA substrate in an attempt to electrically disconnect and isolate arrhythmogenic foci originating from the pulmonary veins (PVs). Multiple catheter technologies for RF have been developed. Catheters may be either cooled or not. Cooling allows for higher and deeper energy delivery with larger lesion formation. Open irrigation cooled-tip RF ablation of AF is associated with less impedance rise, microbubble formation, and esophageal injury when compared with traditional non-cooled ablation catheters. It is also associated with shorter RF delivery time, fluoroscopy, and procedural time.

Understanding the temporal sequence of events of LA structural remodeling (preceding AF ablation) to scar formation (following AF ablation) can prove valuable in determining whether certain patients are more susceptible to recovery of electrical conduction and recurrence of AF. DE-MRI recently has been introduced as a means to visualize this RF-induced scarring post-ablation. These scans can be reconstructed into three-dimensional (3D) recreations of the LA allowing for further analysis and quantification of the LA scar formation following RF ablation.

Objectives:

Primary Objective

• To evaluate the impact of pre-ablation structural remodeling (fibrosis) on scar formation and progression in the LA as assessed by DE-MRI in patients who have undergone successful open irrigated cooled-tipped RF ablation of paroxysmal atrial fibrillation (PAF), using observational, longitudinal data from the University of Utah Comprehensive Arrhythmia Research & Management (CARMA) Center supported AFIB database (approved IRB #20347) over a 12-month follow up period.

Secondary Objectives

* To determine if secondary variables, such as total ablation time, number of lesions, power delivered, and impedance, may play a significant role in catheter induced scar formation.
* To promulgate future research opportunities in the field of AF, particularly with regards to possible early intervention measures that may impact its progression.
* To adapt treatments aimed at patients with AF who are diagnosed at earlier stages.
* To use DE-MRI to further the knowledge and understanding of RF ablation therapy and to better understand the benefits and longitudinal effects of using scar formation to eliminate the fibrotic tissue that conducts the impulses which leads to AF.

ELIGIBILITY:
Inclusion Criteria:

* > 17 years-old and < 90 years-old
* Long-term care for PAF
* Participated in regular clinical follow-ups

Exclusion Criteria:

* Patients who did not receive long-term follow-up care defined as at least 12-months post ablation.
* Women who were pregnant during the time period to be covered by this study.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Forty patients ages 18-89 years, who have had an open irrigation cooled-tipped RF ablation procedure for PAF. Patients must participate in 3-, 6-, and 12-months follow-up post ablation. PAF is defined by >2 documented episodes of AF that terminate spontaneously within 7 days. AF has to be documented by means of electrocardiography, holter monitor, loop recorder, or echocardiography.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nassir F Marrouche, MD, Principal Investigator — University of Utah

REFERENCES:
- [Background] Badger TJ, Oakes RS, Daccarett M, Burgon NS, Akoum N, Fish EN, Blauer JJ, Rao SN, Adjei-Poku Y, Kholmovski EG, Vijayakumar S, Di Bella EV, MacLeod RS, Marrouche NF. Temporal left atrial lesion formation after ablation of atrial fibrillation. Heart Rhythm. 2009 Feb;6(2):161-8. doi: 10.1016/j.hrthm.2008.10.042. Epub 2008 Nov 6. PMID 19187904
- [Background] McGann CJ, Kholmovski EG, Oakes RS, Blauer JJ, Daccarett M, Segerson N, Airey KJ, Akoum N, Fish E, Badger TJ, DiBella EV, Parker D, MacLeod RS, Marrouche NF. New magnetic resonance imaging-based method for defining the extent of left atrial wall injury after the ablation of atrial fibrillation. J Am Coll Cardiol. 2008 Oct 7;52(15):1263-71. doi: 10.1016/j.jacc.2008.05.062. PMID 18926331
- [Background] Marrouche NF, Guenther J, Segerson NM, Daccarett M, Rittger H, Marschang H, Schibgilla V, Schmidt M, Ritscher G, Noelker G, Brachmann J. Randomized comparison between open irrigation technology and intracardiac-echo-guided energy delivery for pulmonary vein antrum isolation: procedural parameters, outcomes, and the effect on esophageal injury. J Cardiovasc Electrophysiol. 2007 Jun;18(6):583-8. doi: 10.1111/j.1540-8167.2007.00879.x. Epub 2007 May 9. PMID 17490437
- [Background] Haissaguerre M, Jais P, Shah DC, Takahashi A, Hocini M, Quiniou G, Garrigue S, Le Mouroux A, Le Metayer P, Clementy J. Spontaneous initiation of atrial fibrillation by ectopic beats originating in the pulmonary veins. N Engl J Med. 1998 Sep 3;339(10):659-66. doi: 10.1056/NEJM199809033391003. PMID 9725923
- [Background] Marrouche NF, Schweikert R, Saliba W, Pavia SV, Martin DO, Dresing T, Cole C, Balaban K, Saad E, Perez-Lugones A, Bash D, Tchou P, Natale A. Use of different catheter ablation technologies for treatment of typical atrial flutter: acute results and long-term follow-up. Pacing Clin Electrophysiol. 2003 Mar;26(3):743-6. doi: 10.1046/j.1460-9592.2003.00126.x. PMID 12698676
- [Result] Oakes RS, Badger TJ, Kholmovski EG, Akoum N, Burgon NS, Fish EN, Blauer JJ, Rao SN, DiBella EV, Segerson NM, Daccarett M, Windfelder J, McGann CJ, Parker D, MacLeod RS, Marrouche NF. Detection and quantification of left atrial structural remodeling with delayed-enhancement magnetic resonance imaging in patients with atrial fibrillation. Circulation. 2009 Apr 7;119(13):1758-67. doi: 10.1161/CIRCULATIONAHA.108.811877. Epub 2009 Mar 23. PMID 19307477

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited based on chart review
Period: Overall Study
Arm/Group | Open Irrigation
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Irrigation
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 26
Age Continuous [Mean (Standard Deviation); unit: years] | 65.2 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Left Atrial (LA) Remodeling Pre-ablation
Description: Utah staging for fibrosis (I - <=5%, II - 5.01%-20.0%, III - 20.01%-35% and IV - >=35.01%)
Time Frame: Once pre-ablation
Measure: Number; unit: participants
Arm/Group | Open Irrigation
Number analyzed (Participants) | 40
participants
  Utah stage 1 | 2
  Utah stage 2 | 31
  Utah stage 3 | 7
  Utah stage 4 | 0
Statistical Analysis 1: Comparison: Open Irrigation; Test type: Superiority or Other; p = 0.48, Regression, Linear; Regression coefficient = 0.13

ADVERSE EVENTS:
Time Frame: This was a retrospective, observational study. Patients were enrolled using chart review. Hence, it did not include collection of adverse events.
Arm/Group | Open Irrigation
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The sample size was too small to see any significant relationship.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No